CLINICAL TRIAL: NCT00401323
Title: A Randomized Phase II-III Multicenter Trial of Docetaxel Plus Cisplatin and Docetaxel Plus 5-FU Versus Cisplatin Plus 5-FU in 1st Line Treatment of Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Taxotere (Docetaxel) in 1st Line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6051; XRP6976G-322
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Head and Neck Neoplasms; Neoplasm Recurrence, Local; Neoplasm Metastasis
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Recurrence, Local; Neoplasm Metastasis | interventions — Docetaxel; Cisplatin; Fluorouracil

ARMS (3):
- docetaxel plus cisplatin (Experimental): Taxotere 75 mg/m², one-hour IV infusion on Day 1 of each 3-week cycle followed by cisplatin 75 mg/m² administered as a 30-minute to 3-hour infusion on Day 1
  Interventions: Drug: docetaxel (XRP6976); Drug: cisplatin
- cisplatin plus 5-FU (Active Comparator): Cisplatin 100 mg/m², 30-minute to 3-hour infusion on Day 1 of each 3-week cycle followed by the continuous infusion of 5-FU 1000 mg/m²/day from Day 1 to Day 5
  Interventions: Drug: cisplatin; Drug: 5-fluorouracil (5-FU)
- docetaxel plus 5-FU (Experimental): Taxotere 85 mg/m², one-hour IV infusion on Day 1 of each 3-week cycle followed by the continuous infusion of 5-FU 750 mg/m²/day from Day 1 to Day 5
  Arm only in the phase II part of the study
  Interventions: Drug: docetaxel (XRP6976); Drug: 5-fluorouracil (5-FU)

INTERVENTIONS:
Drug: docetaxel (XRP6976)
  Other Names: Taxotere
  Arms: docetaxel plus 5-FU; docetaxel plus cisplatin
Drug: cisplatin
  Arms: cisplatin plus 5-FU; docetaxel plus cisplatin
Drug: 5-fluorouracil (5-FU)
  Arms: cisplatin plus 5-FU; docetaxel plus 5-FU

SUMMARY:
The purpose of the study is to compare time to progression and overall survival after treatment with Taxotere plus cisplatin versus cisplatin plus 5-FU (PF treatment group) in the first line treatment of patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically or cytologically documented squamous cell carcinoma of the head and neck (SCCHN) (eligible primary sites: oral cavity, oropharynx, hypopharyx, or larynx) presenting with locally recurrent and/or metastatic disease, with at least 1 unidimensionally or bidimensionally measurable lesion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 1998-01; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
time to progression | up to 5 years

SECONDARY OUTCOMES:
overall survival, overall response rate (complete response + partial response), duration of response, and time to treatment failure | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- sanofi-aventis US, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- sanofi-aventis, Australia, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis, Vienna, Austria
- sanofi-aventis, Belgium, Diegem, Belgium
- Sanofi-Aventis, Rio de Janeiro, Brazil
- sanofi-aventis Canada, Laval, Quebec, Canada
- sanofi-aventis, France, Paris, France
- sanofi-aventis Germany, Berlin, Germany
- sanofi-aventis Greece, Athens, Greece
- Sanofi-Aventis, Basse-Terre, Guadeloupe
- Sanofi-Aventis Hungaria, Budapest, Hungary
- sanofi-aventis Israel, Netanya, Israel
- sanofi-aventis Italy, Milan, Italy
- Sanofi-Aventis, Saint-Denis, Reunion
- Sanofi-Aventis, Moscow, Russia
- sanofi-aventis South Africa, Midrand, South Africa
- Sanofi-Aventis, Madrid, Spain
- sanofi-aventis Switzerland, Geneva, Switzerland
- Sanofi-Aventis, Montevideo, Uruguay